CLINICAL TRIAL: NCT02611726
Title: Effectiveness of Acupuncture Added to Standard Care Vs Standard Care Alone During In-Vitro-Fertilization: A Randomized Controlled Trial
Brief Title: Acupuncture for Symptom Control During Assisted Reproductive Treatments Procedures
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, Max.Cohen, M.D, Bnai Zion Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BnaiZionIVF
Record Dates: First submitted 2015-11-02; First posted 2015-11-23 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Infertility; Pain
MeSH Terms: conditions — Infertility; Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture treatment (Active Comparator): Individualized acupuncture needle insertion according to traditional Chinese and Japanese medicine on top of standard medical care during In-Vitro-Fertilization. Acupuncture needles will be inserted to body surface points following traditional diagnosis (anamnesis, tongue, pulse and abdomen inspection) according to practitioner discretion.
  Interventions: Other: Acupuncture
- Control (No Intervention): Standard medical care during In-Vitro-Fertilization.

INTERVENTIONS:
Other: Acupuncture — Acupuncture
  Arms: Acupuncture treatment

SUMMARY:
Rationale for conducting the experiment: Israel performed IVF treatments since 1980.

Although ART (Advanced Reproductive Treatments) have evolved over the years implantation and pregnancy rates have not met the expectations yet. Success rates of fertility treatments are about 15-18% (clinical pregnancy rates =CPR). As a result additional methods (clinical, technological and complimentary) have been tried to improve the CPR.

In some reviews the effects of acupuncture practice during fertility treatments showed certain benefits, including pain relief and relaxation. Unfortunately those trials were not randomized and lacked methodological rigor.

The aim of this study is to evaluate the effect of acupuncture on pain, anxiety, and CPR of women undergoing IVF as compared to standard care alone.

DETAILED DESCRIPTION:
Women planned for IVF at the investigators' institution will be offered to participate in this trial. Following consent, women will be randomized to acupuncture in addition to standard care OR standard care only according to the working days of the acupuncture practitioner (working alternately three days a week).

After IVF stimulation protocol the patients in the acupuncture group will have three acupuncture treatments: The first will take place right after oocytes retrieval and the second treatment will be right before embryo transfer, and lastly 20-30 minutes after embryo transfer. Patients in the control group will receive standard care only. Patients in both groups will fill out questionnaires regarding expectations from complementary medicine (likert scale no expectation--high expectation), anxiety level (Visual Analogue Scale= VAS) before the procedures, as well as pain assessment (VAS) before and after the IVF procedures. In addition, a general satisfaction questionnaire from the overall care at the IVF unit will be completed at the last visit (likert scale very unsatisfied--highly satisfied). Finally, the physicians will report procedure ease or complexity on a likert scale (very easy-very difficult).

ELIGIBILITY:
Inclusion Criteria:

* Any patient who under going an IVF treatment in the investigators' unit.

Exclusion Criteria:

* Patient who disagree to participate in the study,
* Patient who are undergoing ovulation induction or AID.

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Anxiety before In-Vitro-Fertilization pickup assessed using Visual Analogue Scales (no anxiety 0-10 worst anxiety). | Before and after acupuncture treatments prior to IVF 15 minutes before pickup and 15 minutes after pickup.
  Anxiety will be reported by patients on Visual Analogue Scales (VAS). Mean change in anxiety level will be compared between groups.
Pain level during In-Vitro-Fertilization pickup assessed using Visual Analogue Scale (no pain 0-10 worst pain) | Pain during pickup will be assessed 15 minutes after pickup.
  Pain will be reported by patients on Visual Analogue Scales (VAS). Mean pain level will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Calderon, MD, Study Chair — Deputy CEO, Bnai Zion Medical Center